CLINICAL TRIAL: NCT05035329
Title: Validity and Reliability of Turkish Version of Lower Extremity Functional Scale in Elders
Brief Title: Turkish Version of Lower Extremity Functional Scale in Elders
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Güzin Kara, Principal Investigator, Pamukkale University
Other Study IDs: E-60116787-020-29008
Record Dates: First submitted 2021-08-03; First posted 2021-09-05 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Elders
Keywords: elders; Lower Extremity Functional Scale; validity; reliability; Turkish version

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Outcome measurements — Outcome measurements were applied.

SUMMARY:
This study was conducted in order to analyze the validity and reliability, and psychometric properties of the Turkish version of the Lower Extremity Functional Scale (LEFS-T) in elder adults. The LEFS was translated and cross-culturally adapted to Turkish. Totally 214 elders were included in the study. The LEFS-T, Five-Times-Sit-to-Stand Test (FTSTS), and Falls Efficacy Scale International (FES-I) were applied to all older adults. Item-total correlations of factors and Cronbach alpha internal consistency coefficients were determined to examine the reliability. The relationship between the LEFS-T, FTSTS, and FES-I was analyzed. Exploratory (EFA) and confirmatory factor analysis (CFA) were used for construct validity. Spearman Correlation Analysis was used for concurrent validity. Davis technique was used to calculate the content validity index. Floor and ceiling effect were calculated. It has been concluded that the LEFS-T has good psychometric qualities and can be recommended as a choice of measurement tool to assess self-reported physical functioning in elder adults.

DETAILED DESCRIPTION:
Purpose: This study was conducted in order to analyze the validity and reliability, and psychometric properties of the Turkish version of the Lower Extremity Functional Scale (LEFS-T) in elder adults.

Method: The LEFS was translated and cross-culturally adapted to Turkish. Totally 214 elders were included in the study. The LEFS-T, Five-Times-Sit-to-Stand Test (FTSTS), and Falls Efficacy Scale International (FES-I) were applied to all older adults. Item-total correlations of factors and Cronbach alpha internal consistency coefficients were determined to examine the reliability. The relationship between the LEFS-T, FTSTS, and FES-I was analyzed. Exploratory and confirmatory factor analysis were used for construct validity. Spearman Correlation Analysis was used for concurrent validity. Davis technique was used to calculate the content validity index. Floor and ceiling effect were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years old and older, and ability to speak and read Turkish fluently.

Exclusion Criteria:

* Having neurological, cognitive, and communication problems that can affect the lower extremity functionality severely, and elder adults who cannot answer questionnaires due to inability to understand.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study included 65 years old and elder adults.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2017-10-21 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
Lower Extremity Functional Scale | seven days
  The Lower Extremity Functional Scale was translated and cross-culturally adapted to Turkish. Items are scored as a 5-point Likert Scale (0 = extreme difficulty/ unable to perform an activity, 4 = no difficulty). The highest total score of 80 indicates that the person has a high functional level.
Five-Times-Sit-to-Stand Test | seven days
  The elders were instructed to stand from a standard chair five consecutive times as fast as possible.The duration of the test was recorded in terms of seconds. Less duration means better performance.
Falls Efficacy Scale International | seven days
  The Prevention of Falls Network Europe developed the Falls Efficacy Scale International to assess people's fear of falling during daily living activities. The items score between 1 (not at all concerned) to 4 (very concerned).

CONTACTS AND LOCATIONS:
Overall Officials: Güzin Kara, PhD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Kınıklı/Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Background] Cacchio A, De Blasis E, Necozione S, Rosa F, Riddle DL, di Orio F, De Blasis D, Santilli V. The Italian version of the lower extremity functional scale was reliable, valid, and responsive. J Clin Epidemiol. 2010 May;63(5):550-7. doi: 10.1016/j.jclinepi.2009.08.001. Epub 2009 Nov 12. PMID 19913388